CLINICAL TRIAL: NCT02115646
Title: Fractionated Carbon Dioxide Laser and Burn Scar Contractures: Evaluation of Post-Treatment Scar Function and Appearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shriners Hospitals for Children (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011P001310
Record Dates: First submitted 2013-07-01; First posted 2014-04-16 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Burn Scars
Keywords: burn; scar
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fractionated carbon dioxide laser (Experimental): fractionated carbon dioxide laser
  Interventions: Device: fractionated carbon dioxide laser

INTERVENTIONS:
Device: fractionated carbon dioxide laser — patients will have serial laser treatments
  Other Names: UltraPulse, Lumenis

SUMMARY:
The investigators are studying the appearance and function of burn scars after treatment with fractionated carbon dioxide laser. The investigators hypothesize that the cosmetic appearance and range of motion will improve with treatment.

DETAILED DESCRIPTION:
The primary goal of the study will analyze whether the fractionated carbon dioxide laser can improve other subjective and objective qualities of hypertrophic and/or contracted burn scars with or without involvement of nearby mobile joints.

The investigators hypothesize that fractionated carbon dioxide laser therapy will increase range of motion and improve tissue compliance in all scars overlying a mobile joint that has been limited due to burn scar contracture. In addition, the investigators will evaluate the effect of fractionated carbon dioxide laser therapy on common sequelae of hypertrophic and/or contracted burn scars.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between 5 and 70 years of age with hypertrophic and/or contracted burn scars with or without involvement of mobile joints. The burn scars must have occurred at least 1 year prior to the date of enrollment.
* Having suitable areas of treatment: All wounds in the area of interest must be closed for at least two months, and the scars must be deemed stable for a period of 3 months before initiation of treatment.
* Fitzpatrick skin types I-VI
* Able and willing to comply with all visit, treatment and evaluation schedules and requirements
* Able to understand provide written informed consent
* Women of child-bearing age are required to be using a reliable method of birth control at least three months prior to study enrollment and throughout the course of the study.

Exclusion Criteria:

* Pregnant, intending to become pregnant during the course of the study, less than three months postpartum or less than six weeks after completion of breastfeeding.
* Active tanning, including the use of tanning booths, during the course of the study
* Showing symptoms of hormonal disorders (i.e.: uncontrolled thyroid disease or Polycystic Ovary Syndrome), as per the Investigator's discretion
* Abnormal photosensitivity due to metabolic disorder or due to use of external agents, (drugs, herbs, etc.) within 2 weeks of initial treatment or during the course of the study, except for use of aminolevulinic acid(Levulan®) which requires a washout period of three months
* Prior use of retinoids in treated areas within three months of initial treatment or during the course of the study
* Use of oral isotretinoin (Accutane®) within nine months of initial treatment or during the course of the study. Note: skin must retain its normal degree of moisture prior to treatment
* Prior skin treatment with laser or other devices in the treated area within three months of initial treatment or during the course of the study
* Adverse reactions to compounds of any external agent (e.g., gels, lotions or anesthetic creams) required for use in the study, if no alternative to the said agent exists
* History of collagen vascular disease
* Concurrent inflammatory skin conditions, including, but not limited to, rosacea of any severity
* Active Herpes Simplex at the time of treatment or having experienced more than three episodes of Herpes Simplex eruption within a year of study enrollment
* Multiple dysplastic nevi in area to be treated
* Having a bleeding disorder or taking anticoagulation medications, including heavy use of aspirin, in a manner which does not allow for a minimum 10 day washout period prior to each treatment (as per the patient's physician discretion)
* History of immunosuppression/immune deficiency disorders (including human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS) or use of immunosuppressive medications
* Having any form of active cancer at the time of enrollment and during the course of the study
* Significant concurrent illness, such as uncontrolled diabetes, (i.e., any disease state that in the opinion of the Investigator would interfere with the anesthesia, treatment, or healing process)
* Mentally incompetent, prisoner or evidence of active substance or alcohol abuse
* Any condition which, in the Investigator's opinion, would make it unsafe (for the subject or study personnel) to treat the subject as part of this research study
* If it is determined that the contracture is due to a deeper process involving the muscles, ligaments or bones.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Anderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Shriners Hospital- Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Miletta N, Siwy K, Hivnor C, Clark J, Shofner J, Zurakowski D, Anderson RR, Lee K, Donelan M. Fractional Ablative Laser Therapy is an Effective Treatment for Hypertrophic Burn Scars: A Prospective Study of Objective and Subjective Outcomes. Ann Surg. 2021 Dec 1;274(6):e574-e580. doi: 10.1097/SLA.0000000000003576. PMID 31469749

RESULTS

PARTICIPANT FLOW:
Groups:
- Fractionated CO2 Laser Treatment: Fractionated carbon dioxide laser
  Fractionated carbon dioxide laser: patients received serial fractionated CO2 laser treatments for a total fo 3 treatments.
Period: Overall Study
Arm/Group | Fractionated CO2 Laser Treatment
Started | 29
Completed | 22
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: Subjects with hypertrophic burn scars.
Arm/Group | Fractionated CO2 Laser Treatment
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Scar pigmentation [Mean (Full Range); unit: units on a scale] — This is a measurement of the pigmentation of the scar using a colorimeter device. The scale is rated using a range of 0-100 units, with 100 being the deepest hyperpigmentation, and 0 being no hyperpigmentation.
  units on a scale | 50.93 [13 to 88]
Scar elasticity [Mean (Standard Deviation); unit: units on a scale] — This is the measure of the elasticity of the scar using a Torque-meter. It is measured on a 0-1 unit scale, with 0 being normal skin elasticity and 1 being completely inelastic.
  units on a scale | 0.65 (0.12)
Scar thickness [Mean (Standard Deviation); unit: mm] — This is an ultrasound measurement using the Dermascan Cyberderm to measure the thickness of the scar at baseline in millimeters.
  mm | 3.28 (1.21)
Quality of Life [Mean (Standard Deviation); unit: units on a scale] — The 36-Item Short Form Survey (SF-36) is a validated quality of life measurement tool. It measures 8 health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. It is scored on a 0-100 scale, with 100 being the least bothersome to quality of life.
  units on a scale | 91.25 (8.56)
POSAS [Mean (Standard Deviation); unit: units on a scale] — The Patient and Observer Scar Assessment Scale (POSAS) is a validated scale that measures both the patient assessment and the observer assessment on the quality (height, color, stiffness, thickness, symptoms, relief, surface area) of the scar. Scores range from 0-60, with 60 being the worst quality of scar.
  units on a scale | 27.2 (1.8)

OUTCOME MEASURES:

1. Primary Outcome: Scar Pigmentation, Baseline vs 15-months
Description: Using the colorimeter, will measure change in pigmentation of the scar at the conclusion of the study. This tool measures the pigment in a scar, with a possible range of 0-100, with 100 being the darkest hyperpigmentation, and 0 being no hyperpigmentation.
Time Frame: Baseline and 15 months
Population: All subjects who completed the study (1 baseline visit, 3 fractionated CO2 laser treatments, 1 exit visit) were evaluated.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline: Characteristics of study population at baseline.
- 15-months: Characteristics of study population at conclusion of study.
Arm/Group | Baseline | 15-months
Number analyzed (Participants) | 22 | 22
units on a scale | 50.93 (4.3) | 49.59 (4.1)

2. Primary Outcome: Scar Elasticity, Baseline vs 15-months
Description: This is the measure of the elasticity of the scar using a Torque-meter. It is measured on a 0-1 unit scale, with 0 being normal skin elasticity and 1 being completely inelastic.
Time Frame: Baseline and 15 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | 15-months
Number analyzed (Participants) | 22 | 22
units on a scale | 0.65 (0.12) | 0.49 (0.10)

3. Primary Outcome: Scar Thickness
Description: This is an ultrasound measurement using the Dermascan Cyberderm to measure the thickness of the scar at baseline in millimeters.
Time Frame: Baseline and 15 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Groups:
- 15-months: Characteristics of study population at 15-months
Arm/Group | Baseline | 15-months
Number analyzed (Participants) | 22 | 22
mm | 3.28 (1.21) | 2.58 (1.01)

4. Secondary Outcome: Quality of Life
Description: The 36-Item Short Form Survey (SF-36) is a validated quality of life measurement tool. It measures 8 health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. It is scored on a 0-100 scale, with 100 being the least bothersome to quality of life.
Time Frame: Baseline and 15 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline | 15-months
Number analyzed (Participants) | 22 | 22
units on a scale | 91.25 (8.56) | 97.22 (3.70)

5. Secondary Outcome: POSAS
Description: The Patient and Observer Scar Assessment Scale (POSAS) is a validated scale that measures both the patient assessment and the observer assessment on the quality (height, color, stiffness, thickness, symptoms, relief, surface area) of the scar. Scores range from 0-60, with 60 being the worst quality of scar.
Time Frame: Baseline and 15 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Baseline | 15-months
Number analyzed (Participants) | 22 | 22
units on a scale | 27.2 (1.8) | 15.8 (2.4)

ADVERSE EVENTS:
Arm/Group | Fractionated CO2 Laser Treatment
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes